CLINICAL TRIAL: NCT02390739
Title: Phase I/II Study Administering Peripheral Blood Lymphocytes Transduced With a Murine T-Cell Receptor Recognizing Human Thyroglobulin to Patients With Thyroglobulin Expressing Thyroid Cancer
Brief Title: Administering Peripheral Blood Lymphocytes Transduced With a Murine T-Cell Receptor Recognizing Human Thyroglobulin to People With Thyroglobulin Expressing Thyroid Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 150090; 15-C-0090
Record Dates: First submitted 2015-03-17; First posted 2015-03-18 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2017-03-22

CONDITIONS: Metastatic Thyroid Cancer
Keywords: Immunotherapy; Gene Therapy; Metastatic Cancer
MeSH Terms: conditions — Thyroid Neoplasms; Neoplasm Metastasis | interventions — aldesleukin; fludarabine; Cyclophosphamide

ARMS (1):
- Single Arm (Experimental): All patients will receive a non-myeloablative lymphocyte depleting preparative regimen of cyclophosphamide and fludarabine followed by antithyroglobulin mTCR PBL and aldesleukin.
  Interventions: Drug: Aldesleukin; Drug: Fludarabine; Drug: Cyclophosphamide; Biological: Anti-Thyroglobulin mTCR PBL

INTERVENTIONS:
Drug: Aldesleukin — Aldeskeukin 720,000 IU/kg IV over 15 minutes approximately every eight hours (+/- 1 hour) beginning within 24 hours of cell infusion and continuing for up to 3 days (maximum of 9 doses).
Drug: Fludarabine — Day -7 to -3:Fludarabine 25 mg/m2/day IVPB daily over 30 minutes for 5 days.
Drug: Cyclophosphamide — Days -7 and -6:Cyclophosphamide 60 mg/kg/day X 2 days IV in 250 ml D5W over 1 hour.
Biological: Anti-Thyroglobulin mTCR PBL — On day 0, one to four days after last dose of fludarabine, cells will be infused intravenously (IV) over 20 to 30 minutes.

SUMMARY:
Background

The NCI Surgery Branch has developed an experimental therapy for treating patient with metastatic thyroid cancer that involves taking white blood cells from the patient, growing them in the laboratory in large numbers, genetically modifying these specific cells with a type of virus (retrovirus) to attack only the tumor cells, and then giving the cells back to the patient. This type of therapy is called gene transfer. In this protocol, we are modifying the patient s white blood cells with a retrovirus that has the gene for anti-thyroglobulin incorporated in the retrovirus.

Objectives:

The purpose of this study is to see if these tumor fighting cells (genetically modified cells) that express the receptor for the thyroglobulin molecule on their surface can cause thyroid tumors to shrink and to see if this treatment is safe.

Eligibility:

<TAB>Adults 18 and older with thyroid cancer that has the thyroglobulin molecule on tumor surfaces

Design:

<TAB>Work up stage: Patients will be seen as an outpatient at the NIH clinical Center and undergo a history and physical examination, scans, x-rays, lab tests, and other tests as needed

<TAB>Leukapheresis: If the patients meet all of the requirements for the study they will undergo leukapheresis to obtain white blood cells to make the anti- thyroglobulin cells. {Leukapheresis is a common procedure, which removes only the white blood cells from the patient.}

<TAB>Treatment: Once their cells have grown, the patients will be admitted to the hospital for the conditioning chemotherapy, the anti-thyroglobulin cells and aldesleukin. They will stay in the hospital for about 4 weeks for the treatment.

Follow up:

Patients will return to the clinic for a physical exam, review of side effects, lab tests, and scans about every 1-3 months for the first year, and then every 6 months to 1 year as long as their tumors are shrinking. Follow up visits take up to 2 days.

DETAILED DESCRIPTION:
Background:

* We generated a murine T-cell receptor (mTCR) that recognizes human thyroglobulin (hTG) in the context of HLA-A0201 and constructed a single retroviral vector that contains its alpha and beta chains and will confer hTG recognition to HLA-A0201+ PBL on transduction.
* In co-cultures with HLA-A0201+, hTG+ target cells, anti-TG mTCR transduced T cells secrete significant amounts of IFN- >= with high specificity.

Objectives:

Primary objectives:

* To determine the safety of administering PBL transduced with this anti-TG mTCR in concert with preparative lymphodepletion and high dose interleukin-2 (IL-2; aldesleukin).
* Determine if these mTCR-transduced PBL can mediate the regression of TG-expressing tumors.

Eligibility:

Patients who are HLA-A*0201 positive and 18 years of age or older must have

-Advanced TG-expressing thyroid cancer (including those with bone-only disease) which has progressed after surgery (if indicated) and radioiodine ablation

Patients may not have:

-Contraindications for high dose aldesleukin administration.

Design:

* PBMC obtained by leukapheresis will be cultured in the presence of anti-CD3 (OKT3) and aldesleukin in order to stimulate T-cell growth.
* Transduction is initiated by exposure of these cells to retroviral vector supernatant containing replication-incompetent virus encoding the anti-TG mTCR.
* All patients will receive a non-myeloablative lymphocyte depleting preparative regimen of cyclophosphamide and fludarabine.
* On day 0 patients will receive their PBL transduced with the anti-TG mTCR and then begin high dose aldesleukin.
* A complete evaluation of evaluable lesions will be conducted approximately 4-6 weeks after treatment.
* The study will be conducted using a Phase I/II optimal design.
* The objective will be to determine if the combination of high dose aldesleukin, lymphocyte depleting chemotherapy, and anti-TG mTCR-gene engineered lymphocytes is able to be associated with a clinical response rate that can rule out 5% (p0=0.05) in favor of a modest 20% PR + CR rate (p1=0.20).
* A total of up to 68 patients may be required; approximately 25 patients in the phase I portion of the study and 43 (41, plus an allowance of up to 2 non-evaluable) patients in the phase II portion of the study.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Unresectable thyroid cancer expressing TG as assessed by one of the following methods: RT-PCR on tumor tissue, or by immunohistochemistry of resected tissue.
  2. Recurrent/metastatic radioiodine refractory disease that has progressed within the past 6 months with at least 1 lesion increasing by 0.5cm in diameter or with increasing bone metastases.
  3. Confirmation of diagnosis of thyroid cancer by the Laboratory of Pathology of the NCI.
  4. PET avid disease with SUV >5.
  5. Patients must have previously received standard systemic therapy for advanced thyroid cancer (to include radioactive iodine for iodine-avid tumors and surgery (if indicated)) and have been either non-responders (progressive disease) or have recurred.
  6. Patients with 3 or fewer brain metastases that are less than 1 cm in diameter and asymptomatic are eligible. Lesions that have been treated with stereotactic radiosurgery must be clinically stable for 1 month after treatment for the patient to be eligible.
  7. Greater than or equal to 18 years of age and less than or equal to 70 years of age.
  8. Willing to sign a durable power of attorney
  9. Able to understand and sign the Informed Consent Document
  10. Clinical performance status of ECOG 0 or 1
  11. Life expectancy of greater than three months
  12. Patients must be HLA-A*0201 positive
  13. Patients of both genders must be willing to practice birth control from the time of enrollment on this study and for up to four months after treatment.
  14. Serology:
* Seronegative for HIV antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune-competence and thus be less responsive to the experimental treatment and more susceptible to its toxicities.)
* Seronegative for hepatitis B antigen, and seronegative for hepatitis C antibody. If hepatitis C antibody test is positive, then patient must be tested for the presence of antigen by RT-PCR and be HCV RNA negative.

  o. Women of child-bearing potential must have a negative pregnancy test because of the potentially dangerous effects of the treatment on the fetus.

  p. Hematology
* Absolute neutrophil count greater than 1000/mm3 without the support of filgrastim
* WBC less than or equal to 3000/mm3
* Platelet count greater than or equal to 100,000/mm3
* Hemoglobin greater than 8.0 g/dl

  q. Chemistry:
* Serum ALT/AST less than or equal to to 2.5 times the upper limit of normal
* Serum creatinine less than or equal to to 1.6 mg/dl
* Total bilirubin less than or equal to to 1.5 mg/dl, except in patients with Gilbert s Syndrome who must have a total bilirubin less than 3.0 mg/dl.

  r. More than four weeks must have elapsed since any prior systemic therapy at the time the patient receives the preparative regimen, and patients toxicities must have recovered to a grade 1 or less (except for toxicities such as alopecia or vitiligo).

Note: Patients may have undergone minor surgical procedures within the past 3 weeks, as long as all toxicities have recovered to grade 1 or less.

EXCLUSION CRITERIA:

1. Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the treatment on the fetus or infant.
2. Any form of primary immunodeficiency (such as Severe Combined

   Immunodeficiency Disease).
3. Active systemic infections (e.g. : requiring anti-infective treatment), coagulation disorders or other major medical illnesses of the cardiovascular, respiratory or immune system, myocardial infarction, cardiac arrhythmias, obstructive or restrictive pulmonary disease.
4. Concurrent opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities).
5. Concurrent systemic steroid therapy.
6. History of severe immediate hypersensitivity reaction to cyclophosphamide or fludarabine.
7. History of coronary revascularization or ischemic symptoms
8. Documented LVEF of less than or equal to 45%. Testing is required in patients with:

   * Clinically significant atrial and/or ventricular arrhythmias including but not limited to: atrial fibrillation, ventricular tachycardia, second or third degree heart block
   * Age greater than or equal to 60 years old

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-03-02; Primary Completion 2017-03-22 (Actual); Study Completion 2017-03-22 (Actual)

PRIMARY OUTCOMES:
Determine a safe dose of administration and determine if this approach will result in an objective tumor regression. | Approximately 4 years

CONTACTS AND LOCATIONS:
Overall Officials: James C Yang, M.D., Principal Investigator — National Cancer Institute (NCI)

REFERENCES:
- [Background] Siegel R, Naishadham D, Jemal A. Cancer statistics, 2013. CA Cancer J Clin. 2013 Jan;63(1):11-30. doi: 10.3322/caac.21166. Epub 2013 Jan 17. PMID 23335087
- [Background] Castro MR, Bergert ER, Goellner JR, Hay ID, Morris JC. Immunohistochemical analysis of sodium iodide symporter expression in metastatic differentiated thyroid cancer: correlation with radioiodine uptake. J Clin Endocrinol Metab. 2001 Nov;86(11):5627-32. doi: 10.1210/jcem.86.11.8048. PMID 11701745
- [Background] Droz JP, Schlumberger M, Rougier P, Ghosn M, Gardet P, Parmentier C. Chemotherapy in metastatic nonanaplastic thyroid cancer: experience at the Institut Gustave-Roussy. Tumori. 1990 Oct 31;76(5):480-3. doi: 10.1177/030089169007600513. PMID 2256195